CLINICAL TRIAL: NCT03788317
Title: Integrated Botulinum Toxin for Improved Sitting Balance in Children With Cerebral Palsy: Body Functions to Activity and Participation
Brief Title: Improved Sitting Balance: Body Functions to Participation
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Nigar Dursun, Professor, Kocaeli University
Other Study IDs: KU GOKAEK 2018/358
Record Dates: First submitted 2018-12-25; First posted 2018-12-27 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy, Botulinum Toxin A, Participation
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Botulinum toxin type A — Injections to hypertonic muscles
  Other Names: Botox, Dysport

SUMMARY:
The aim of this study is to evaluate the changes in activity and participation domains of International Classification of Functioning, Disability and Health (ICF) in children with cerebral palsy (CP) who received integrated Botulinum Toxin-A (BoNT-A) injections into the lower limb(s) with a treatment goal of improved sitting balance.

DETAILED DESCRIPTION:
Postural problems play a substantial role in activities of daily living in children with CP having Gross Motor Function Classification System (GMFCS) levels IV or V. Improvement in sitting balance may positively effect the performance and caregiving of vital tasks of daily life in these children and may furtherly improve the quality of life of both the child and family. BoNT-A is an important treatment in children with CP because it is safe in young children and allows combined treatment. In the current literature its efficacy on body functions and structures by hypertonia management is well known. However there is inconclusive evidence for improvement in activity and participation domains of ICF with BoNT-A. CP is a very heterogenous population and in most of the studies the inclusion criteria do not adress level of underlying motor control and the primary efficacy assessment methods were usually chosen to cover hypertonia. Besides generally the efficacy endpoints were so soon to detect changes in activity or participation domains of ICF. Lack of association of rehabilitation programs is another important concern for the current clinical studies.

In this present study a well defined subpopulation of CP children having GMFCS levels of IV or V who each received integrated BoNT-A treatment with a primary goal of improved sitting balance will be recruited to identify the probable changes in activity and participation domains of ICF as well as changes in quality of life of the family and the child.

ELIGIBILITY:
Inclusion Criteria:

* All children with a diagnosis of cerebral palsy with respect to Rosenbaum criteria
* Gross Motor Functional Classification Scale level of IV-V
* Being scheduled for BoNT-A treatment to lower extremity
* Primary goal of treatment selected as improved sitting balance

Exclusion Criteria:

* Severe cognitive or behavioural problems
* Severe dystonia

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children diagnosis of cerebral palsy with respect to Rosenbaum criteria having received BoNT-A injections to lower limb(s) as well as an integrated treatment approach
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
The Child and Adolescent Scale of Participation (CASP) | 20 weeks
  Participation measurement The CASP consists of 20 ordinal-scaled items and four subsections: 1) Home Participation 2) Community Participation 3) School Participation and 4) Home and Community Living Activities The 20 items are rated on a four-point scale: Age Expected (Full participation) to Unable.
The Caregiver Priorities & Child Health Index of Life with Disabilities (CPCHILD) | 20 weeks
  Health Related Quality of Life measurement The CPCHILD© Questionnaire measures the caregiver's perspective about the child's health status, comfort, wellbeing, functional abilities and ease of caregiving. It is a useful proxy measure of health related quality of life of children with severe disabilities.
  Basic Scoring Procedure Scores for each domain and for the total survey are standardized and range from 0 (worse) to 100 (best).

SECONDARY OUTCOMES:
Goal Assessment Scale (GAS) | 20 weeks
  Functional goal attainment measurement GAS 5-Point Rating Scale Score Predicted Attainment
  (-2)Less than expected outcome
  (-1) Expected outcome after intervention
  (0)Much less than expected outcome
  (+1) Greater than expected outcome
  (+2) Much greater than expected outcome

OTHER OUTCOMES:
Gross Motor Function Classification System (GMFCS) | 20 weeks
  Motor Development The gross motor skills (e.g. sitting and walking) of children and young people with cerebral palsy can be categorised into 5 different levels from I to V using a tool called GMFCS.
Mean change from baseline Modified Ashworth Scale (MAS) | 20 weeks
  Tone measurement Scoring 0= No increase muscle tone; 1= Slight increase ın muscle tone, manifested by a catch and release or by minimal resislance at the end of the range of motion when the affected part (s) is moved in flexion or extension;
  1+=Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM; 2 =More marked increase in muscle tone through most of the ROM, but affected part (s) easily moved; 3 =Considerable increase in muscle tone, passive movement difficult; 4 =Affected part (s) rigid in flexion or extension.
Mean change from baseline angle of catch (XV3) Tardieu scale | 20 weeks
  Spasticity measurement Degree of anle of catch is measured baseline and after treatment to define the change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nigar Dursun, Study Director — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nguyen L, Di Rezze B, Mesterman R, Rosenbaum P, Gorter JW. Effects of Botulinum Toxin Treatment in Nonambulatory Children and Adolescents With Cerebral Palsy: Understanding Parents' Perspectives. J Child Neurol. 2018 Oct;33(11):724-733. doi: 10.1177/0883073818786567. Epub 2018 Jul 24. PMID 30039731
- [Background] Nguyen L, Mesterman R, Gorter JW. Development of an inventory of goals using the International Classification of Functioning, Disability and Health in a population of non-ambulatory children and adolescents with cerebral palsy treated with botulinum toxin A. BMC Pediatr. 2018 Jan 4;18(1):1. doi: 10.1186/s12887-017-0974-x. PMID 29301539
- [Background] Delgado MR, Tilton A, Russman B, Benavides O, Bonikowski M, Carranza J, Dabrowski E, Dursun N, Gormley M, Jozwiak M, Matthews D, Maciag-Tymecka I, Unlu E, Pham E, Tse A, Picaut P. AbobotulinumtoxinA for Equinus Foot Deformity in Cerebral Palsy: A Randomized Controlled Trial. Pediatrics. 2016 Feb;137(2):e20152830. doi: 10.1542/peds.2015-2830. Epub 2016 Jan 26. PMID 26812925
- [Background] Dursun N, Gokbel T, Akarsu M, Dursun E. Randomized Controlled Trial on Effectiveness of Intermittent Serial Casting on Spastic Equinus Foot in Children with Cerebral Palsy After Botulinum Toxin-A Treatment. Am J Phys Med Rehabil. 2017 Apr;96(4):221-225. doi: 10.1097/PHM.0000000000000627. PMID 27631386
- [Background] Reid SM, Carlin JB, Reddihough DS. Using the Gross Motor Function Classification System to describe patterns of motor severity in cerebral palsy. Dev Med Child Neurol. 2011 Nov;53(11):1007-12. doi: 10.1111/j.1469-8749.2011.04044.x. PMID 22014320